CLINICAL TRIAL: NCT03811535
Title: A Trial Comparing the Effect and Safety of Once Weekly Dosing of Somapacitan With Daily Norditropin® in Children With Growth Hormone Deficiency
Brief Title: A Research Study in Children With a Low Level of Hormone to Grow. Treatment is Somapacitan Once a Week Compared to Norditropin® Once a Day (REAL4)
Acronym: REAL4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4263; U1111-1207-9691 (Other: World Health Organization (WHO)); 2018-000231-27 (Other: European Medicines Agency (EudraCT)); JapicCTI-194773 (Registry Identifier: JAPIC (Japan))
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Growth Hormone Deficiency in Children
MeSH Terms: interventions — somapacitan; Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: Participants will receive either somapacitan once weekly or Norditropin® once daily for 52 weeks (main trial period). All participants completing the main trial period will receive somapacitan weekly for 3 years (extension trial period).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Somapacitan weekly (Experimental): Participants will receive somapacitan weekly for 52 weeks (main trial period). Participants completing the main trial period in both the treatment arms ('Somapacitan weekly' and 'Norditropin® daily') will receive somapacitan weekly for 3 years (extension trial period).
  Interventions: Drug: Somapacitan
- Norditropin® daily (Active Comparator): Participants will receive Norditropin® daily for 52 weeks (main trial period).
  Interventions: Drug: Norditropin®

INTERVENTIONS:
Drug: Somapacitan — Somapacitan will be administered subcutaneously (s.c.; under the skin) once weekly by PDS290 pen-injector. Somapacitan can be injected any time during the once weekly dosing day. The dose will be calculated based on the subject's current body weight.
  Arms: Somapacitan weekly
Drug: Norditropin® — Norditropin® will be administered s.c. once daily by FlexPro® pen-injector. Norditropin® should be injected daily in the evening. The dose will be calculated based on the subject's current body weight.
  Arms: Norditropin® daily

SUMMARY:
The study compares 2 medicines for children who do not have enough hormone to grow: somapacitan given once a week (a new medicine) and Norditropin® given once a day (the medicine doctors can already prescribe). Researchers will test to see how well somapacitan works. The study will also test if somapacitan is safe. Participants will either get somapacitan or Norditropin® - which treatment participants get, is decided by chance. Both participants and the study doctor will know which treatment participants get. The study will last for 4 years. Participants will attend 19 clinic visits and have 1 phone call with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal children: a) Boys: Age more than or equal to 2 years and 26 weeks and less than 11.0 years at screening. Testis volume less than 4 ml. b) Girls: Age more than or equal to 2 years and 26 weeks and less than 10.0 years at screening. Tanner stage 1 for breast development (no palpable glandular breast tissue)
* Confirmed diagnosis of growth hormone deficiency determined by two different growth hormone stimulation tests performed within 12 months prior to randomisation, defined as a peak growth hormone level of less than or equal to 10.0 ng/ml using the World Health Organisation (WHO) International Somatropin 98/574 standard
* Impaired height defined as at least 2.0 standard deviations below the mean height for chronological age and gender at screening according to the standards of Center for Disease Control and Prevention
* Impaired height velocity, defined as annualised height velocity below the 25th percentile for chronological age and gender according to the standards of Prader calculated over a time span of minimum 6 months and maximum 18 months prior to screening
* Insulin-like Growth Factor-I (IGF-I) less than -1.0 SDS at screening, compared to age and gender normalized range measured at central laboratory
* No prior exposure to growth hormone therapy or IGF-I treatment

Exclusion Criteria:

* Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with standing height measurements
* Current inflammatory diseases requiring systemic corticosteroid treatment for longer than 2 consecutive weeks within the last 3 months prior to screening
* Children requiring inhaled glucocorticoid therapy at a dose of greater than 400 μg/day of inhaled budesonide or equivalents for longer than 4 consecutive weeks within the last 12 months prior to screening
* Diagnosis of attention deficit hyperactivity disorder
* Concomitant administration of other treatments that may have an effect on growth, e.g. but not limited to methylphenidate for treatment of attention deficit hyperactivity disorder
* Prior history or presence of malignancy including intracranial tumours

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (135):
- United States (27):
  - Univ of AL at Birmingham_BRM, Birmingham, Alabama
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hosp Of Orange, Orange, California
  - Sutter Valley Med Fdt Ped Endo, Sacramento, California
  - Rocky Mt Ped and Endo, Centennial, Colorado
  - Ped Endo Assoc PC-G.V, Greenwood Village, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - A.I. duPont Hospital for Children/Nemours, Wilmington, Delaware
  - Pediatric Endocrine & Wellness Center, Aventura, Florida
  - Van Meter Pediatric Endo PC, Atlanta, Georgia
  - Riley Hospital For Children, Indianapolis, Indiana
  - University OF Iowa, Iowa City, Iowa
  - Univ of Minnesota M.C.H., Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota
  - Children's Mercy Clinics, Kansas City, Missouri
  - The Docs, Las Vegas, Nevada
  - Goryeb Children's Hospital, Morristown, New Jersey
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - NYU Langone Hospital-LI, Mineola, New York
  - WakeMed Childn Endo-Dbt_Raleig, Raleigh, North Carolina
  - CCHMC_Cinc, Cincinnati, Ohio
  - Univ Oklahoma Sci Ctr OK City, Oklahoma City, Oklahoma
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
  - Dell Children's Medical Center, Austin, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - MultiCare Inst for Res & Innov, Tacoma, Washington
- Algeria (3):
  - CHU Bab El Oued Pediatrics Dept, Algiers
  - Endo and Diab Dept El Oued, Algiers
  - endocrino-diabetology department, Hospital IBN BADIS., Constantine
- Austria (4):
  - Med. Univ. Graz -Klinische Abteilung f. Allgemeine Pädiatrie, Graz
  - LKH Salzburg- Univ. Klinik f. Kinder- und Jugendheilkunde, Salzburg
  - LKH St. Poelten, Kinder-und Jugendheilkunde, Sankt Pölten
  - Salzkammergut-Klinikum Vöcklabruck, Vöcklabruck
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Mntrl Chldrn Hsptl PedEndoMUHC, Montreal, Quebec
- Rigshospitalet Klinik for Vækst og Reproduktion Afsnit 5064, Copenhagen Ø, Denmark
- Estonia (2):
  - Tallinn Children's Hospital, Tallinn
  - Tartu University Hospital Children's Clinic, Tartu
- France (8):
  - Centre Hospitalier Universitaire D'Angers-2, Angers
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Pellegrin, Bordeaux
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - Hopital de Bicetre_Le Kremlin-Bicetre, Le Kremlin-Bicêtre
  - Assistance Publique Hopitaux de Marseille-Hopital de La Timone-2, Marseille
  - Hopital de La Timone, Marseille Cédex 05
  - Ap-Hp-Hopital Necker-2, Paris
  - HOPITAL DES ENFANTS-HOPITAL PAULE DE VIGUIER - Pharmacie, Toulouse
- Germany (4):
  - Endokrinologikum Frankfurt, Frankfurt am Main
  - Auf der Bult Medizinisches Versorgungszentrum Hannover, Hanover
  - Uniklinik Tübingen - Kinder- und Jugendmedizin, Tübingen
  - Uniklinik Ulm - Dt. Zentrum für Kinder- und Jugendgesundheit (DZKJ), Ulm
- Hungary (2):
  - Észak-Közép-budai Centrum, Szent János Kórház és Szakrendelő, Budapest
  - Szegedi Tudományegyetem Gyermekgyógyászati Klinika, Szeged
- India (3):
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Dehli, New Delhi
- CHI Crumlin Dept of Endocrinology, Dublin, Ireland
- Israel (4):
  - Rambam MC - Department of Pediatrics A, Haifa
  - Meir MC - Department of Paediatrics, Kfar Saba
  - Schneider MC - Endrocrinology and Diabetes, Petah Tikva
  - Shamir MC - Pediatric and Adolescents Endocrinology unit, Ẕerifin
- Italy (4):
  - IRCCS Meyer Firenze, Florence
  - Ospedale Pediatrico Gaslini, Genova
  - Ospedale Maggiore Policlinico UO Endocrinologia Diabetolgia, Milan
  - Ospedale Pediatrico Bambino Gesu, Roma
- Japan (23):
  - Kurume University Hospital, Pediatrics, Fukuoka
  - Fukuoka Children's Hospital_Endocrinology and Metabolism, Fukuoka-shi, Fukuoka
  - National Hospital Organization FUKUYAMA MEDICAL CENTER, Fukuyama-shi, Hiroshima
  - Fukuyama City Hospital_Department of Pediatrics, Fukuyama-shi, Hiroshima
  - Kanagawa Children's Medical Center, Dev. Endo and Metabo, Kanagawa
  - Hyogo Prefectual Kobe Children's Hospital Dept. Metab & endo, Kobe-shi, Hyogo
  - Univ.HP, Kyoto Pref Univ of Medicine, Dept. of Pediatrics, Kyoto
  - Ibaraki Children's Hospital_General Pediatrics, Mito, Ibaraki
  - Nara Prefecture General Medical Center_ Nara-shi, Nara, Nara-shi, Nara
  - Niigata University Medical & Dental Hospital_Pediatrics, Niigata-shi, Niigata
  - Aichi Children's Health and Medical Center, Obu-shi, Aichi
  - Okayama Medical Center_Cardiology, Okayama-shi, Okayama
  - Osaka City General Hospital, Pediatric Endocrinology and Me, Osaka
  - Osaka Women's and Children's Hospital, Osaka
  - Saitama Children's Medical Center, Endocrinorogy&Metabolism, Saitama-shi, Saitama
  - Hamamatsu Univ. School of Medicine Hospital, Pediatrics, Shizuoka
  - Osaka University Hospital_Pediatrics, Suita-shi, Osaka
  - Institute of Science Tokyo Hospital_Pediatrics, Tokyo
  - KOUJIYA Kodomo Clinic, Tokyo
  - National Center for Child Health and Dev, Endo and Metabo, Tokyo
  - Tanaka Growth Clinic, Tokyo
  - Keio University Hospital, Pediatrics, Tokyo
  - Tokyo Metropolitan Children's Medical Center_Endo and Metab, Tokyo
- Children's Clinical University Hospital, Riga, Latvia
- Haukeland Universitetssykehus, Barneklinikken, Bergen, Norway
- Poland (3):
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - SPSK nr 1 im Prof. T Sokolowskiego, Szczecin
  - Instytut ''Pomnik - Centrum Zdrowia Dziecka'', Warsaw
- Russia (8):
  - Republic Children's Hospital of Ministry of Health of Udmurt, Izhevsk
  - Setchenov First Moscow State Medical University, Moscow
  - RMAPE, Moscow
  - Children's clinical city hospital #1, Novosibirsk
  - FSBEI of Higher Education "Rostov State Medical University", Rostov-on-Don
  - SPSBHI City Children out-patient clinic #44, Saint Petersburg
  - Samara Regional Children Clinical Hospital n.a. N.N. Ivanova, Samara
  - Siberian State Medical University, Tomsk
- Serbia (5):
  - University Clinical Centre Nis, Niš, RS
  - University Children's Hospital Tirsova, Belgrade
  - Institute for Mother and Child Health Care of Serbia, Belgrade
  - University Clinical Centre Kragujevac, Kragujevac
  - Institute for Health Care of Children and Adolescents, Novi Sad
- University Children's Hospital, Ljubljana, Slovenia
- South Korea (11):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center_Seoul, Seoul
- Spain (2):
  - Hospital Clínico de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Sant Joan de Déu, Esplugues Llobregat(Barcelona)
- Switzerland (3):
  - Universitäts-Kinderspital beider Basel, Basel
  - Med. Kinder- und Poliklinik, Bern
  - Kinderspital Endokrinologie, Zürich, Zurich
- Thailand (2):
  - King Chulalongkorn Memorial hospital_Ped-Endocrinology, Bangkok
  - Phramongkutklao Hospital_Ped-Endo_Pediatrics, Bangkok
- Ukraine (3):
  - Kharkiv Regional Children's Clinical Hospital - Endocrinological department, Kharkiv
  - Komisarenko Institute of Endocrinology and Metabolism of NAMSU - Department of paediatric endocrine pathology, Kyiv
  - Vinnytsia Regional Clinical Endocrinological Centre - Therapeutic department #2, Vinnytsia
- United Kingdom (7):
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - Hull Royal Infirmary, Hull
  - Alder Hey Children's Hospital, Liverpool
  - Royal London Hospital_London, London
  - Royal Manchester Children's Hospital, Manchester
  - St George's Hospital, Tooting
  - St Georges Hospital, Tooting

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com

REFERENCES:
- [Derived] Miller BS, Blair JC, Rasmussen MH, Frystyk J, Lemminger AK, Maniatis A, Mori J, Bottcher V, Kim HS, Polak M, Horikawa R. Efficacy, safety, and insulin-like growth factor I of weekly somapacitan in children with growth hormone deficiency: 3-year results from REAL4. Eur J Endocrinol. 2025 Apr 30;192(5):651-661. doi: 10.1093/ejendo/lvaf096. PMID 40400262
- [Derived] Mori J, Ohata Y, Fujisawa Y, Sato Y, Rohrich S, Rasmussen MH, Bang RB, Horikawa R. Effective growth hormone replacement with once-weekly somapacitan in Japanese children with growth hormone deficiency: Results from REAL4, a phase 3 clinical trial. Clin Endocrinol (Oxf). 2024 Apr;100(4):389-398. doi: 10.1111/cen.15025. Epub 2024 Feb 18. PMID 38368603
- [Derived] Miller BS, Blair JC, Rasmussen MH, Maniatis A, Mori J, Bottcher V, Kim HS, Bang RB, Polak M, Horikawa R. Effective GH Replacement With Somapacitan in Children With GHD: REAL4 2-year Results and After Switch From Daily GH. J Clin Endocrinol Metab. 2023 Nov 17;108(12):3090-3099. doi: 10.1210/clinem/dgad394. PMID 37406251
- [Derived] Miller BS, Blair JC, Rasmussen MH, Maniatis A, Kildemoes RJ, Mori J, Polak M, Bang RB, Bottcher V, Stagi S, Horikawa R. Weekly Somapacitan is Effective and Well Tolerated in Children With GH Deficiency: The Randomized Phase 3 REAL4 Trial. J Clin Endocrinol Metab. 2022 Nov 25;107(12):3378-3388. doi: 10.1210/clinem/dgac513. PMID 36062966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 86 sites in 20 countries as follows (number of sites that screened participants/ number of sites that randomized participants): Austria (2/1); Canada (1/1); Denmark (1/0); France (4/4); Germany (3/2); Hungary (1/0); India (3/3); Israel (4/4); Italy (3/2); Japan (17/14); Korea (8/6); Latvia (1/1); Poland (1/1); Russia (8/8); Serbia (5/3); Slovenia (1/1); Spain (2/2); Switzerland (1/1); Thailand (2/2); Ukraine (3/3); United Kingdom (5/5); United States (23/22).
Pre-assignment Details: Data reported based on the main part of the trial i.e. up to week 52.
Groups:
- Norditropin: Participants received 0.034 milligrams/kilogram (mg/kg) norditropin subcutaneously (s.c.; under the skin) by FlexPro pen-injector once daily for 52 weeks (main trial period). Participants completing the main trial period will receive 0.16 mg/kg somapacitan once weekly for 3 years (extension period).
- Somapacitan: Participants received 0.16 mg/kg somapacitan s.c. once weekly by PDS290 pen-injector for 52 weeks (main trial period). Participants completing the main trial period will receive 0.16 mg/kg somapacitan once weekly for 3 years (extension period).
Period: Overall Study
Arm/Group | Norditropin | Somapacitan
Started | 68 | 132
Completed | 68 | 132
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Norditropin | Somapacitan | Total
Number analyzed (Participants) | 68 | 132 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.43 (2.42) | 6.38 (2.23) | 6.40 (2.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 33 | 51
  Male | 50 | 99 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 63 | 119 | 182
  Unknown or Not Reported | 4 | 9 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 36 | 78 | 114
  Race: Asian | 28 | 46 | 74
  Race: Black or African American | 1 | 0 | 1
  Race: Other | 0 | 1 | 1
  Race: Not reported | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity: In-trial Observation Period
Description: Height velocity (HV) was derived from height measurements taken at baseline and Week 52 visit as: HV = (height at 52 weeks visit - height at baseline)/(time from baseline to 52 weeks visit in years). Data is reported for 'in-trial' observation period. In-trial observation period: from first administration and up until visit 7 or last trial contact, whichever comes first.
Time Frame: From baseline (week 0) to visit 7 (week 52)
Population: Full analysis set included all randomized participants.
Measure: Mean (Standard Deviation); unit: centimeters per year (cm/year)
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 68 | 132
centimeters per year (cm/year) | 11.8 (2.9) | 11.2 (2.5)
Statistical Analysis 1: Comparison: Norditropin vs Somapacitan; Height velocity at week 52 was analyzed using an analysis of covariance model with treatment, gender, age group, region, growth hormone (GH) peak group and gender by age group by region interaction term as factors, and baseline height as covariate; Test type: Non-Inferiority — The pre-specified non-inferiority margin was -1.8 cm/year; ANCOVA; Treatment difference = -0.5, 95% CI 2-sided [-1.1 to 0.2]

2. Primary Outcome: Height Velocity: On-treatment Observation Period
Description: Height velocity was derived from height measurements taken at baseline and Week 52 visit as: HV = (height at 52 weeks visit - height at baseline)/(time from baseline to 52 weeks visit in years). Data is reported for 'on-treatment' observation period. On-treatment observation period: from first administration and up until last trial contact, visit 7 or 14 days after last administration, whichever comes first.
Time Frame: From baseline (week 0) to visit 7 (week 52)
Population: Full analysis set included all randomized participants. Overall Number of Participants Analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 68 | 131
cm/year | 11.8 (2.9) | 11.2 (2.5)
Statistical Analysis 1: Comparison: Norditropin vs Somapacitan; Height velocity at 52 weeks was analyzed using a mixed model for repeated measurements, with treatment, gender, age group, region, GH peak group and gender by age group by region interaction terms as factors and baseline height as a covariate, all nested within week as a factor; Test type: Non-Inferiority — The pre-specified non-inferiority margin was -1.8 cm/year; Mixed Models Analysis; Treatment difference = -0.5, 95% CI 2-sided [-1.1 to 0.2]

3. Secondary Outcome: Change in Bone Age
Description: Change from baseline (week -2) in bone age at week 52 is presented. X-ray images of left hand and wrist for bone age assessment according to the Greulich and Pyle atlas were taken. In-trial observation period: from first administration and up until visit 7 or last trial contact, whichever comes first.
Time Frame: Baseline (week -2), week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 68 | 131
Years | 1.28 (0.76) | 1.13 (0.78)

4. Secondary Outcome: Change in Height Standard Deviation Score (HSDS)
Description: Change from baseline (week 0) in HSDS at week 52 is presented. HSDS was derived using Centre for Disease Control and Prevention (CDC) standards. The range for HSDS was -10 to +10. Negative scores indicated a height below the mean height for a child with the same age and gender, whereas positive scores indicated a height above the mean height for a child with the same age and gender. Positive value in change from baseline in HSDS indicated that HSDS was better than baseline HSDS. In-trial observation period: from first administration and up until visit 7 or last trial contact, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: Full analysis set included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 68 | 132
Score on a scale | 1.37 (0.69) | 1.21 (0.54)

5. Secondary Outcome: Change in Height Velocity Standard Deviation Score (HV SDS)
Description: Change from baseline (week 0) in HV SDS at week 52 is presented. HV SDS was calculated using the formula: HV SDS = (height velocity - mean)/standard deviation (SD), where height velocity was the height velocity variable measured, mean and SD of height velocity by gender and age for the reference population. The range for HV SDS was -10 to +10. Negative scores indicated a height velocity below the mean height velocity for a child with the same age and gender, whereas positive scores indicated a height velocity above the mean height velocity for a child with the same age and gender. Positive value in change from baseline in HV SDS indicated that HV SDS was better than baseline HV SDS. In-trial observation period: from first administration and up until visit 7 or last trial contact, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: Full analysis set included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 68 | 132
Score on a scale | 8.97 (4.38) | 7.97 (3.36)

6. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) at Week 52
Description: Change from baseline (week -2) in FPG at week 52 is presented.
Time Frame: Baseline (week -2), week 52
Population: Safety analysis set included all randomized participants exposed to at least one dose of randomized treatment. Overall Number of Participants Analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 66 | 124
Millimoles per liter (mmol/L) | 0.255 (0.790) | 0.083 (0.567)

7. Secondary Outcome: Change in FPG at Week 104
Time Frame: Baseline (week -2), week 104
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Change in FPG at Week 156
Time Frame: Baseline (week -2), week 156
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Change in FPG at Week 208
Time Frame: Baseline (week -2), week 208
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Change in Homeostatic Model Assessment Steady State Beta Cell Function (HOMA-B) at Week 52
Description: Change from baseline (week -2) in HOMA-B at week 52 is presented. HOMA-B is a measure of the beta cell function and was calculated as follows: HOMA-B = (20 * fasting insulin (picomoles per liter [pmol/L]) * 1/6(microunit per milliliter [µU/mL]))/ FPG(mmol/L)-3.5). Negative change from baseline in HOMA-B indicated a worse outcome.
Time Frame: Baseline (week -2), week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of HOMA-B
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 58 | 111
Percentage of HOMA-B | 69.24 (81.59) | 37.71 (59.25)

11. Secondary Outcome: Change in HOMA-B at Week 104
Time Frame: Baseline (week -2), week 104
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: Change in HOMA-B at Week 156
Time Frame: Baseline (week -2), week 156
Reporting Status: Not Posted, anticipated posting 2025-12

13. Secondary Outcome: Change in HOMA-B at Week 208
Time Frame: Baseline (week -2), week 208
Reporting Status: Not Posted, anticipated posting 2025-12

14. Secondary Outcome: Change in Homeostatic Model Assessment Insulin Resistance (HOMA-IR) at Week 52
Description: Change from baseline (week -2) in HOMA-IR at week 52 is presented. HOMA-IR is an evaluation of the insulin resistance and was calculated as HOMA-IR = fasting insulin (pmol/L) * 1/6(µU/mL) * FPG(mmol/L) / 22.5. Positive change from baseline in HOMA-IR indicated a worse outcome.
Time Frame: Baseline (week -2), week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of HOMA-IR
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 60 | 114
Percentage of HOMA-IR | 1.03 (1.12) | 0.60 (1.13)

15. Secondary Outcome: Change in HOMA-IR at Week 104
Time Frame: Baseline (week -2), week 104
Reporting Status: Not Posted, anticipated posting 2025-12

16. Secondary Outcome: Change in HOMA-IR at Week 156
Time Frame: Baseline (week -2), week 156
Reporting Status: Not Posted, anticipated posting 2025-12

17. Secondary Outcome: Change in HOMA-IR at Week 208
Time Frame: Baseline (week -2), week 208
Reporting Status: Not Posted, anticipated posting 2025-12

18. Secondary Outcome: Change in Glycated Haemoglobin (HbA1c) at Week 52
Description: Change from baseline (week -2) in HbA1c at week 52 is presented.
Time Frame: Baseline (week -2), week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 68 | 130
Percentage of HbA1c | 0.11 (0.26) | 0.09 (0.22)

19. Secondary Outcome: Change in HbA1c at Week 104
Time Frame: Baseline (week -2), week 104
Reporting Status: Not Posted, anticipated posting 2025-12

20. Secondary Outcome: Change in HbA1c at Week 156
Time Frame: Baseline (week -2), week 156
Reporting Status: Not Posted, anticipated posting 2025-12

21. Secondary Outcome: Change in HbA1c at Week 208
Time Frame: Baseline (week -2), week 208
Reporting Status: Not Posted, anticipated posting 2025-12

22. Secondary Outcome: Change in Insulin-like Growth Factor I (IGF-I) Standard Deviation Score (SDS) at Week 52
Description: Change from baseline (week 0) in IGF-I SDS at week 52 is presented. The range for IGF-I SDS was from -10 to +10. Negative scores indicated a IGF-I below the mean IGF-I for a child with the same age and gender, whereas positive scores indicated a IGF-I above the mean IGF-I for a child with the same age and gender. For participants with low IGF-I SDS at baseline, a positive change from baseline in IGF-I SDS indicated a better outcome. Data is reported for 'in-trial' observation period. In-trial observation period: from first administration and up until visit 7 or last trial contact, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 67 | 132
Score on a scale | 2.41 (1.09) | 2.32 (1.27)

23. Secondary Outcome: Change in IGF-I SDS at Week 104
Time Frame: Baseline (week 0), week 104
Reporting Status: Not Posted, anticipated posting 2025-12

24. Secondary Outcome: Change in IGF-I SDS at Week 156
Time Frame: Baseline (week 0), week 156
Reporting Status: Not Posted, anticipated posting 2025-12

25. Secondary Outcome: Change in IGF-I SDS at Week 208
Time Frame: Baseline (week 0), week 208
Reporting Status: Not Posted, anticipated posting 2025-12

26. Secondary Outcome: Change in Insulin-like Growth Factor Binding Protein 3 (IGFBP-3) Standard Deviation Score (SDS) at Week 52
Description: Change from baseline (week 0) in IGFBP-3 SDS at week 52 is presented. The range for IGFBP-3 SDS was from -10 to +10. Negative scores indicated a IGFBP-3 below the mean IGFBP-3 for a child with the same age and gender, whereas positive scores indicated a IGFBP-3 above the mean IGFBP-3 for a child with the same age and gender. For participants with low IGFBP-3 SDS at baseline, a positive change from baseline in IGFBP-3 SDS indicated a better outcome. Data is reported for 'in-trial' observation period. In-trial observation period: from first administration and up until visit 7 or last trial contact, whichever comes first.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin | Somapacitan
Number analyzed (Participants) | 67 | 132
Score on a scale | 1.68 (1.02) | 1.58 (0.92)

27. Secondary Outcome: Change in IGFBP-3 SDS at Week 104
Time Frame: Baseline (week 0), week 104
Reporting Status: Not Posted, anticipated posting 2025-12

28. Secondary Outcome: Change in IGFBP-3 SDS at Week 156
Time Frame: Baseline (week 0), week 156
Reporting Status: Not Posted, anticipated posting 2025-12

29. Secondary Outcome: Change in IGFBP-3 SDS at Week 208
Time Frame: Baseline (week 0), week 208
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: From week -2 up to week 52
Description: Safety analysis set included all randomized participants exposed to at least one dose of randomized treatment.
Arm/Group | Norditropin | Somapacitan
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/132
Serious Adverse Events (participants affected / at risk) | 2/68 | 6/132
Other Adverse Events (participants affected / at risk) | 22/68 | 46/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (N=68) | Somapacitan (N=132)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin (N=68) | Somapacitan (N=132)
Bronchitis (Infections and infestations) | 5 (5) | 4 (6)
Headache (Nervous system disorders) | 6 (11) | 16 (22)
Nasopharyngitis (Infections and infestations) | 7 (13) | 15 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 12 (17)
Pyrexia (General disorders) | 7 (12) | 10 (14)
Vomiting (Gastrointestinal disorders) | 4 (6) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT03811535/Prot_SAP_000.pdf